CLINICAL TRIAL: NCT05797766
Title: Efficacy of Fluid Distribution Timetable on the Treatment Adherence of End-Stage Renal Disease Patient: A Randomized Controlled Trial
Brief Title: Efficacy Trial of Fluid Distribution Timetable
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Santo Tomas (Other)
Collaborators: University of Santo Tomas Hospital (Unknown)
Responsible Party: Principal Investigator, Joshua Nathaniel Ellano, Principal Investigator, University of Santo Tomas
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: REC-2022-08-095-RN
Record Dates: First submitted 2023-02-28; First posted 2023-04-04 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: End-stage Renal Disease
Keywords: End-stage Renal Disease; Fluid Distribution Timetable; Thirst; Interdialytic weight; Nephrology Nursing; Hemodialysis
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): The fluid distribution timetable as defined by Mina et al. (2019) is a scheduled distribution of predetermined amounts of fluid intake daily depicted in a 5x6 table. The timetable has three major columns. The first column has six-time points of a day with a four-hour interval. The second column, which was divided into four sub-columns, reflects the percentage of fluid allotment for food, activities, medication, and thirst encounters. The percentage of fluid allocation was computed based on the patient's prescribed fluid restriction, usual time of food intake per day, usual level of activity, time of medication intake, and common time they encounter thirst for a day. The third column indicates the converted percentage of fluid allotment into milliliters.
  Interventions: Behavioral: Fluid Distribution Timetable
- Control (No Intervention): Standard care that consists of 10 to 15 minutes of face-to-face health teaching of their treatment regimen including management of medication, vascular access, dietary and fluid, and hemodialysis schedule.

INTERVENTIONS:
Behavioral: Fluid Distribution Timetable — a scheduled distribution of predetermined amounts of fluid intake daily depicted in a 5x6 table. The timetable has three major columns. The first column has six-time points of a day with a four-hour interval. The second column, which was divided into four sub-columns, reflects the percentage of fluid allotment for food, activities, medication, and thirst encounters. The percentage of fluid allocation was computed based on the patient's prescribed fluid restriction, usual time of food intake per day, usual level of activity, time of medication intake, and common time they encounter thirst for a day. The third column indicates the converted percentage of fluid allotment into milliliters.
  Arms: Treatment

SUMMARY:
Nonadherence to fluid restriction is a significant issue among hemodialysis patients globally, with numerous adverse health outcomes. These outcomes include increased intradialytic weight gain, acid-base and electrolyte imbalances, and decreased mental health. This study aimed to determine the effects of a fluid distribution timetable on adherence to fluid restriction among patients with end-stage renal disease undergoing hemodialysis. The study utilized a single-blind, randomized-controlled efficacy trial design. Selected ESRD patients undergoing hemodialysis are then randomized using computer-generated sequences of randomly permuted blocks stratified according to sex to receive the intervention or the control group. Adherence to fluid restriction was measured using the dialysis thirst inventory and intradialytic weight gain. The variables were computed using One-way Repeated Measures Multivariate Analysis of Variance and Multivariate Analysis of Covariance. Secondary outcomes included baseline patient demographic profile and was compared according to group allocation. Both group were followed up for four weeks, assessing the outcome measures during the third hemodialysis session for each week

DETAILED DESCRIPTION:
Chronic Kidney Disease (CKD), a condition wherein the kidney is damaged and cannot filter blood properly (National Institute of Diabetes and Digestive and Kidney Diseases, 2019), if left untreated, end-stage renal disease (ESRD) otherwise known as kidney failure occurs. CKD has been recognized as one of the major public health problems globally and has an estimated prevalence of 13.4% of the total population and ESRD has an estimate between 4.902 million to 7.083 million cases. According to the CKD Health Policy Model, it is projected that there would be an increase of 16.7% cases of CKD in adults in the year 2030.

Hemodialysis is a maintenance management form of renal replacement therapy. It is a treatment to filter the excess fluid and blood wastes by using a special filter that is considered as an artificial kidney. However, hemodialysis alone is not a treatment for this disease, with the help of fluid restriction and change of dietary prescription the quality of life of the patient may significantly improve.

In the perspective of hemodialysis patients, adherence to dietary regimens and fluid restrictions is a great challenge due to the burden of constant choices about food and drink, the adaptation to complex eating patterns, existing cultural practices, and the competing demands of the chronic disease and comorbidities.

Adherence to fluid restriction is a major problem among hemodialysis patients around the world and persists to be a clinical concern in nephrology care. and a clinical problem in nephrology care. Nonadherence to fluid restriction as defined by the National Kidney Foundation is gaining an intradialytic weight of more than 5.7% of their weight post hemodialysis session. Nonadherence to fluid restriction are found to have numerous health-related problems, an increased intradialytic weight gain, acid-base and electrolyte imbalances, and a decrease in mental health. Other than themselves, the hemodialysis patient must also consider the burden of their home caregivers such as the management of family costs, the maintenance of physical and psychological health, the provision of care, the assumption of multiple roles, and the communication of expectations are challenges as a caregiver.

This study is a single-blind, single center, randomized-controlled trial that utilized data collection triangulation to assess the efficacy and feasibility of a nursing intervention that will promote treatment adherence to fluid restriction among hemodialysis patients in a private tertiary level institution in Manila, Philippines.

Sample size computation using G*Power 3.1.7 showed that a sample size of 40 respondents is necessary to achieve a power of 80%, attrition rate of 20%, partial η2 of 0.41, effect size of 0.79 and significance level of 5% (two-tailed). A group allocation of 1:1 was used in five data collection timeframes. The participating patients was allocated randomly into two groups, the intervention, and the control group, using a computer-generated sequence of random permuted blocks. The randomization was stratified according to the participants' sex and was done by an independent statistician. The groupings was not be disclosed to the participants and the unit's personnel in the duration of the study but was be disclosed once the study is done.

Upon consenting, the participants were then divided into two groups using stratified, permuted block randomization. The control group received standard care that consists of 10 to 15 minutes of face-to-face health teaching of their treatment regimen including management of medication, vascular access, dietary and fluid, and hemodialysis schedule. The intervention group received a combination of standard care and the intervention, the fluid distribution timetable. The fluid distribution timetable is a scheduled distribution of predetermined amounts of fluid intake daily depicted in a 5x6 table. The timetable has three major columns. The first column has six-time points of a day with a four-hour interval. The second column, which was divided into four sub-columns, reflects the percentage of fluid allotment for food, activities, medication, and thirst encounters. The percentage of fluid allocation was computed based on the patient's prescribed fluid restriction, usual time of food intake per day, usual level of activity, time of medication intake, and common time they encounter thirst for a day. The third column indicates the converted percentage of fluid allotment into milliliters. The researcher shall provide a 210 ml glass for accuracy and uniformity of measurement of fluid intake at home. The predetermined fluid restriction was determined by the participant's nephrologist. The trained staff nurses was able to teach the intervention to the participant and their primary care provider. The trained nurses answered any questions and queries of the participant or the primary care provider until they understand the intervention fully. If there are questions that the trained nurses cannot answer, the trained staff nurse shall inform the researcher and be answered as soon as possible. The researcher provided multiple copies of the fluid distribution table for each participant in the intervention group. The participants was observed for one month and follow up with their fluid distribution timetable every last day of their hemodialysis for the week and shall be collected by the researcher.

The prerecorded video used for training may also be used for the patient's queries and may also be a guide at home. If the patient has difficulty in understanding the terms that the intervention uses, the researcher may explain the intervention in layman's terms for better understanding. If there is an existing language barrier, the researcher may explain the intervention in the Filipino language. The veracity of the participants can be verified in their intradialytic weight gain in between their previous hemodialysis weight gain and their current pre-hemodialysis weight gain. To eliminate threats to internal validity, the researcher randomized all consented participants upon acquiring informed consent and divided them into two evenly distributed groups, the control and intervention group to eliminate selection bias. The control group is formed to eliminate the threat to history and maturation. To eliminate the threat to temporal ambiguity, the researcher gathered the data of baseline thirst scores and interdialytic weight of all participants. In the event that the participant is unable to attend their scheduled hemodialysis session, the researcher may adjust their schedule as long as they have their hemodialysis three times per week and if they fail to commit to this condition, the participant shall be removed from the study.

Adherence to fluid restriction was measured by utilizing two indicators, thirst and intradialytic weight gain, and was compared using One-way Repeated Measures Multivariate Analysis of Variance and Multivariate Analysis of Covariance. The thirst was measured using a standardized tool, the dialysis thirst inventory, which was self reported by the participants. The intradialytic weight weight gain was computed by determining the difference of the current pre-hemodialysis session weight and the previous post hemodialysis weight. Secondary outcomes included the baseline demographic profile and were compared according to treatment allocation. Both groups were followed up fort four weeks, assessing the outcome measures on the third hemodialysis session of the week

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with End-stage renal disease
* Oliguric (urine output of less than 20ml/ hr)
* Aged 40 - 70 years old
* Had been on dialysis for at least 6 months
* Is alert and oriented
* With scheduled for hemodialysis thrice a week.

Exclusion Criteria:

* Pregnant patients
* Has a history or overt mental illness
* Patients with congestive heart failure

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-01-18 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2023-05-05 (Actual)

PRIMARY OUTCOMES:
Perceived Thirst Score | 4 Weeks
  The Dialysis Thirst Inventory (DTI) measured perceived thirst among the participants. It is a 7-item questionnaire answered on 5-point Likert scale, with scores ranging from 7 to 35 and higher scores indicating higher thirst. No cut-off score is present for the questionnaire; however, higher scores are interpreted as higher perceived thirst.
Intradialytic Weight Gain | 4 Weeks
  It is the net increase in body weight from previous post-dialysis weight measured in kilograms

SECONDARY OUTCOMES:
Age | Week 1
  The age of the respondents in years at the time of participation in the study
Sex | Week 1
  The biological gender of the respondent
Educational Attainment | Week 1
  The highest educational attainment of the respondent at the time of participation of the study
Edema Status | Week 1
  The edema or third space fluid of the respondent at the time of participation of the study
Ultrafiltration Goal | Week 1
  The ultrafiltration goal is categorized by met or unmet of the set ultrafiltration rate of the respondent

CONTACTS AND LOCATIONS:
Locations (1):
- University of Santo Tomas Hospital, Manila, Philippines

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF